CLINICAL TRIAL: NCT00314067
Title: Comprehensive Quality Management in Out-patient Care for Alcohol-related Disorders (AQAH). Transfer and Dissemination Into Routine Practice
Brief Title: Evaluation of Case Management to Improve the Outpatient Care of Alcohol-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BMBF-01EB0412
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2008-06

CONDITIONS: Alcohol-related Disorders
Keywords: Quality of Health Care; Primary Health Care; Education; E-Learning; Alcohol-related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Ethanol; Primary Health Care

ARMS (3):
- 1 (Experimental)
  Interventions: Procedure: Online Comprehensive Quality Management System (CQM) of alcohol-related disorders in primary care; Procedure: Physician training
- 2 (Experimental)
  Interventions: Procedure: Online Comprehensive Quality Management System (CQM) of alcohol-related disorders in primary care; Procedure: Physician training; Procedure: Practice team training
- 3 (Active Comparator)
  Interventions: Procedure: Online Comprehensive Quality Management System (CQM) of alcohol-related disorders in primary care

INTERVENTIONS:
Procedure: Online Comprehensive Quality Management System (CQM) of alcohol-related disorders in primary care
Procedure: Physician training
  Arms: 1; 2
Procedure: Practice team training
  Arms: 2

SUMMARY:
The purpose of this study is to disseminate and transfer the comprehensive quality management interventions (CQM) for alcohol-related disorders in primary care developed during the first funding phase into routine care. The two steps are (1) to optimize the CQM approach and (2) to investigate the dissemination and transfer into routine care in a randomized controlled trial.

DETAILED DESCRIPTION:
In the first funding phase the project AQAH ("Ambulantes Qualitätsmanagement alkoholbezogener Störungen in der hausärztlichen Praxis"-"comprehensive quality management for alcohol-related disorders in primary care") systematically investigated three issues: (1) the outpatient care system and evidence-base for screening, diagnosis and treatment was examined; it developed (2) a comprehensive quality management system (CQM) consisting of documentation material, a pathway of care and evidence-based practice guidelines; (3) the effects of the CQM on the detection and treatment of alcohol-related disorders were investigated in a randomized controlled pre-post design and the results show positive effects of the CQM. In the second funding phase (a 3 year bi-center project) the purpose is now to disseminate and transfer the CQM into routine care. The two steps are (1) to optimize the CQM approach and (2) to investigate the dissemination and transfer into routine care in a randomized trial. (1) The paper-based AQAH-practice guidelines are transformed into an interactive electronic version with online patient documentation and evaluation, decision support measures as well as links to specialists and an e-learning tool. (2) After pilot testing in the AQAH-study-networks, an active transfer to the greater regions of Südbaden and Südwürttemberg will be performed in a parallel group cluster randomized controlled trial with GP practices as unit of randomization. Outcome data will be collected concerning the acceptance of the system and the quality of care delivered.

Comparison(s): (1) Use of the interactive electronic version of the CQM for alcohol-related disorders with a special training for general practitioners, compared to (2) use of the CQM with additional education for the whole practice team and organizational re-structuring advice, compared to (3) a control group who uses the CMQ without any special training.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner
* Possibility to use broad-band internet

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-07; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Acceptance of the CQM-system: Number of actively participating practices
Adherence to the system: relative numbers of screened, documented and followed-up patients

SECONDARY OUTCOMES:
Quality of care provided: Patients that are adequately treated and followed-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin Härter, Prof. Dr. Dr., Principal Investigator — Freiburg University Hospital, Dept. of Psychiatry and Psychotherapy; Michael Berner, Dr., Principal Investigator — Freiburg University Hospital, Dept. of Psychiatry and Psychotherapy; Daniela Ruf, Dipl. Psych., Study Chair — Freiburg University Hospital, Dept. of Psychiatry and Psychotherapy; Götz Mundle, PD Dr., Study Chair — Oberbergklinik, Hornberg and University Hospital for Psychiatry and Psychotherapy, Tübingen; Monika Lohmann, Dipl. Psych., Study Chair — University Hospital for Psychiatry and Psychotherapy, Tübingen
Locations (2):
- Germany (2):
  - Freiburg University Hospital, Dept. of Psychiatry and Psychotherapy, Freiburg im Breisgau
  - University Hospital for Psychiatry and Psychotherapy, Tübingen, Tübingen

REFERENCES:
- [Background] Harter M, Bermejo I, Kratz S, Schneider F. [Continuing education and quality management measures for the implementation of clinical practice guidelines]. Z Arztl Fortbild Qualitatssich. 2003 Nov;97 Suppl 4:67-73. German. PMID 14710670
- [Background] Mänz C, Berner M, Lorenz G, Härter M, Bermejo I, Berger M, Buchkremer G, Mundle G. Projekt AQAH: Ambulantes Qualitätsmanagement alkoholbezogener Störungen beim Hausarzt. Suchtmedizin 5(1): 1-8, 2003.
- [Background] Mänz C, Berner M, Härter M, Lorenz G, Mundle G. Akzeptieren Patienten Screening-Fragebögen für alkoholbezogene Störungen? Nervenarzt 74(2): 261, 2003.
- [Background] Harter M, Bermejo I, Schneider F, Gaebel W, Niebling W, Berger M. [Comprehensive ambulatory care quality management for patients with depressive disorders]. Z Arztl Fortbild Qualitatssich. 2003 Nov;97 Suppl 4:9-15. German. PMID 14710664
- [Background] Berner MM, Habbig S, Harter M. [Quality of guidelines for the treatment of alcohol related disorders -- a systematic review and content analysis]. Fortschr Neurol Psychiatr. 2004 Dec;72(12):696-704. doi: 10.1055/s-2004-830097. German. PMID 15580534
- [Background] Berner M, Mundle G, Lorenz G, Härter M. Möglichkeiten der Frühintervention bei alkoholbezogenen Störungen in der hausärztlichen Praxis. Suchttherapie 5: 70-75, 2004.
- [Background] Berner MM, Zeidler C, Kriston L, Mundle G, Lorenz G, Harter M. [Diagnostic and treatment approaches to alcohol-related disorders]. Fortschr Neurol Psychiatr. 2006 Mar;74(3):157-64. doi: 10.1055/s-2005-870949. German. PMID 16528639
- [Background] Berner MM, Bentele M, Kriston L, Manz C, Clement HW, Harter M, Mundle G. DOVER and QUVER-new marker combinations to detect and monitor at-risk drinking. Alcohol Clin Exp Res. 2006 Aug;30(8):1372-80. doi: 10.1111/j.1530-0277.2006.00163.x. PMID 16899040
- [Derived] Ruf D, Berner M, Kriston L, Lohmann M, Mundle G, Lorenz G, Niebling W, Harter M. Cluster-randomized controlled trial of dissemination strategies of an online quality improvement programme for alcohol-related disorders. Alcohol Alcohol. 2010 Jan-Feb;45(1):70-8. doi: 10.1093/alcalc/agp079. Epub 2009 Nov 4. PMID 19889887